CLINICAL TRIAL: NCT02836743
Title: Effect of Slow-release Melatonin (Circadin®) Therapy on Idiopathic REM Sleep Behavior Disorder: a Pilot Study
Brief Title: Effect of Slow-release Melatonin (Circadin®) Therapy on Idiopathic RBD: a Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Young Jung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1505-084-673
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: REM Sleep Behavior Disorder
Keywords: REM sleep behavior disorder; Melatonin
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Circadin 2mg (Experimental): low-dose (2mg) slow-release melatonin for 1 month.
  Interventions: Drug: Circadin
- Circadin 6mg (Experimental): high-dose (6mg) slow-release melatonin for 1 month.
  Interventions: Drug: Circadin
- Placebo (Placebo Comparator): Administer placebo pills with identical morphology
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Circadin — Slow-release melatonin
  Other Names: slow-release melatonin
  Arms: Circadin 2mg; Circadin 6mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate effect of slow-release melatonin (Circadin) on REM sleep behavior disorder.

DETAILED DESCRIPTION:
Investigators planned to administer low (2mg) and high (6mg) dose slow-release melatonin and the placebo for 4 weeks and evaluate Clinical Global Impression scale, RBD questionnaire, PSQI, Epworth sleepiness scale, and quality of life questionnaire (SF-36v2) before and after the treatment along with possible side effects and drug compliance.

ELIGIBILITY:
Inclusion Criteria:

* REM sleep behavior disorder according to ICSD-3 criteria
* No cognitive deficit or symptom of Parkinsonism
* Those with written consent.

Exclusion Criteria:

* who took medication (ex. clonazepam) for REM sleep behavior disorder
* with degenerative neurologic disorder (ex. Parkinson's disease, Multiple System Atrophy, Lewy-body dementia, etc.)
* who took medication that can affect REM sleep behavior disorder (anti-depressant: SSRI, TCA, MAO-inhibitor)
* who is unable to answer questionnaires
* who have hypersensitive reaction to medications
* Pregnant women or breastfeeding
* who are diagnosed with other parasomnia disorder
* with severe medical disorder (severe liver failure, respiratory failure, heart failure, malignant tumor, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Clinical Global Impression scale | baseline and 4 weeks
Changes in RBDQ-HK score (RBD questionnaire-HK) | Baseline and 4 weeks

SECONDARY OUTCOMES:
Sleep quality questionnaire | after taking the treatment for 4 weeks
  PSQI
Sleepiness questionnaire | after taking the treatment for 4 weeks
  Epworth sleepiness scale
Quality of life questionnaire | after taking the treatment for 4 weeks
  SF-36 version 2.
Changes in Dream enactment behavior frequency described in sleep diary | Baseline and 4 weeks
Drug adverse effect | 4 weeks
  adverse events and reason for drug withdrawal

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Takeuchi N, Uchimura N, Hashizume Y, Mukai M, Etoh Y, Yamamoto K, Kotorii T, Ohshima H, Ohshima M, Maeda H. Melatonin therapy for REM sleep behavior disorder. Psychiatry Clin Neurosci. 2001 Jun;55(3):267-9. doi: 10.1046/j.1440-1819.2001.00854.x. PMID 11422870
- [Background] Kunz D, Bes F. Melatonin as a therapy in REM sleep behavior disorder patients: an open-labeled pilot study on the possible influence of melatonin on REM-sleep regulation. Mov Disord. 1999 May;14(3):507-11. doi: 10.1002/1531-8257(199905)14:33.0.co;2-8. PMID 10348479
- [Background] Boeve BF, Silber MH, Ferman TJ. Melatonin for treatment of REM sleep behavior disorder in neurologic disorders: results in 14 patients. Sleep Med. 2003 Jul;4(4):281-4. doi: 10.1016/s1389-9457(03)00072-8. PMID 14592300
- [Background] Kunz D, Mahlberg R. A two-part, double-blind, placebo-controlled trial of exogenous melatonin in REM sleep behaviour disorder. J Sleep Res. 2010 Dec;19(4):591-6. doi: 10.1111/j.1365-2869.2010.00848.x. PMID 20561180